CLINICAL TRIAL: NCT06205576
Title: A Post Market Clinical Study to Evaluate the Safety and Efficacy of the Acotec Drug-coated Balloon for the Treatment of the Obstructive Lesions in the Native Arteriovenous Dialysis Fistuae(AVF)
Brief Title: ACOART AVF RENEW: A Post Market Clinical Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acotec Scientific Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACOART AVF RENEW
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Stenosis of Native Hemodialysis Arteriovenous Fistulas

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DCB catheter (Experimental): Using DCB catheter for the treatment of subjects with a de novo or non-stented restenotic obstructive lesion located in the native arteriovenous dialysis fistulae.
  Interventions: Device: DCB catheter

INTERVENTIONS:
Device: DCB catheter — Trade name of DCB catheter：Acoart Orchid＆Dhalia

SUMMARY:
The objective of this prospective，multi-center，single arm study is to obtain further data on the safety and performance of the Acotec Orchid＆Dhalia Drug-coated Balloon catheters for the treatment of for the obstructive lesions in the native Arteriovenous Dialysis Fistulae (AVF).

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥18 and ≤85 years of age
* The target AV fistula has undergone successful dialysis for at least 1 time
* Patient has a de novo and/or non-stented restenotic lesion located in the outflow vein（Arteries and Central Vein are excluded）
* Patient has a de novo and/or non-stented restenotic lesion（≥50% stenosis）and at least one of the following occurs：

  * The physical examination was abnormal
  * Significant increase in dynamic venous pressure
  * Blood flow decreased significantly
* Patient has a target lesion or a tandem lesion that is ≤ 100 mm in length
* Patient underwent successful crossing of the target lesion with the guide wire and pre-dilatation with a PTA balloon defined as:

  * Residual stenosis of ≤ 30% AND
  * Absence of a flow limiting dissection (Grade ≥C) or perforation
* Patient provides written informed consent prior to enrollment in the study

Exclusion Criteria:

* Women who are breastfeeding, pregnant, or are intending to become pregnant, or men intending to father children
* Dialysis access is located in the lower extremity
* More than one lesion
* Patient with hemodynamically significant central venous stenoses
* Patient has presence of a stent located in the target AV access circuit
* Patient has undergone prior intervention of access site within 30 days of index procedure
* Patient with target AVF or access circuit which previously had or currently has a plan to surgery
* Patient who cannot receive recommended antiplatelet and/or anticoagulant therapy
* Patients undergoing immunotherapy or suspected/confirmed vasculitis
* Patients with a history of coagulation dysfunction, thrombocytopenic purpura or RH-negative blood type
* Patient has an infected AV access or systemic infection
* Patient has a life expectancy of <24 months
* Patient is anticipating a kidney transplant or with anticipated conversion to peritoneal dialysis
* Patient has a co-morbid condition that, in the judgment of the Investigator, may cause him/her to be non-compliant with the protocol or confound the data interpretation
* Patient is enrolled in another investigational drug, device, or biologic study and has not completed the primary endpoint, or was previously enrolled in this study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Primary Patency Rate | 6 months
  Defined as freedom from clinically-driven target lesion revascularization (CD-TLR) or access circuit thrombosis measured.
Serious Adverse Event Rate | 30 days
  Defined as the Serious Adverse Event (SAE) rate involving the AV access circuit.

SECONDARY OUTCOMES:
Target Lesion Primary Patency Rate | 12 months，24 months
  Defined as freedom from CD-TLR or access thrombosis occurring in the target lesion post-procedure.
All-cause mortality Rate | 24 months
  All-cause mortality post procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Haidian Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No